CLINICAL TRIAL: NCT06621186
Title: Construction of an in Vitro Intestinal Microbial Ecological Simulation System for Obese People
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0953
Record Dates: First submitted 2024-09-29; First posted 2024-10-01 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-09

CONDITIONS: Obese Subjects

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention measures — No intervention measures

SUMMARY:
About 2.6 billion people ( about 40 % of the world 's population ) are affected by overweight or obesity. The prevalence of overweight and obesity in Chinese adults has exceeded 50 %, and the prevalence is still on the rise.The gut microbiota is regarded as an endocrine organ and participates in energy balance. Diet changes can disrupt the relationship between the microbiota and the host, leading to metabolic diseases.Although human studies provide important information, there are limitations, such as the entry of complex gastrointestinal environment limiting components, the lack of dynamic microbial process information, and the uncertainty of drug side effects. In vitro methods can solve these problems, allowing dynamic sampling, standardized operation, high repeatability, and evaluation of potential toxins and pathogens. In vitro models are widely used to evaluate the effects on the human colon microbiome and to predict in vivo results.Based on the above research background, this study aims to collect fecal samples from obese people to construct an in vitro intestinal microbial ecological simulation system. This will lay an experimental foundation for further exploring the effect of specific nutrient intervention on the composition and function of gut microbiota in obese people.

ELIGIBILITY:
Inclusion Criteria:

* Screening in the physical examination population who intend to retain fecal samples in the physical examination center of our hospital. BMI ≥ 28, age range from 18 to 30.

Exclusion Criteria:

* Previous history of intestinal disease, history of hypertension, diabetes, coronary heart disease and other chronic diseases, history of important organ disease or surgery, history of malignant tumor disease.
* He had a history of heavy smoking and alcohol abuse.
* In the past 6 months, she took antibiotics.
* Weight loss measures in the past 6 months, including but not limited to dieting, physical exercise, probiotic intervention and other medications.
* Subjects and their families who disagreed with the study protocol.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: samples in the physical examination center of our hospital. BMI ≥ 28, age range from 18 to 30.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
intestinal microflora | 2025.10
  Construction of simulated intestinal microflora ecosystem

CONTACTS AND LOCATIONS:
Overall Officials: daren Liu, MD, PhD, Study Chair — Chief Physician
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No